CLINICAL TRIAL: NCT07367477
Title: HORIZONTAL VERSUS VERTICAL UPPER EXTREMITY PERFORMANCE ON HAND SKILLS AND TRUNK CONTROL IN BILATERAL CEREBRAL PALSY
Brief Title: Horizontal Versus Vertical Upper Extremity Function in Bilateral Cerebral Palsy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Raghda Gamal Ateya Abd-Elbary (Other)
Responsible Party: Sponsor-Investigator, Raghda Gamal Ateya Abd-Elbary, Physical Therapy Specialist, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/004404
Record Dates: First submitted 2026-01-18; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-02

CONDITIONS: Bilateral Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Active Comparator): Children in this group will receive a designed occupational therapy (OT) program to improvement hand skills conducted on a horizontal surface.
  Interventions: Procedure: a designed occupational therapy (OT) program to improvement hand skills conducted on a horizontal surface.
- Group (B) (Experimental): Children in this group will receive the same designed OT program given to group (A) conducted on a vertical surface.
  Interventions: Procedure: a designed occupational therapy program to improvement hand skills conducted on a vertical surface.

INTERVENTIONS:
Procedure: a designed occupational therapy program to improvement hand skills conducted on a vertical surface. — The treatment session will be started by the following exercises for 30 minutes as preparation for hand skill training and the second part of the session will be exercises facilitating fine motor skills a vertical surface for one hour, Three sessions per week will last for 90 minutes, for successive Three months.
  Arms: Group (B)
Procedure: a designed occupational therapy (OT) program to improvement hand skills conducted on a horizontal surface. — The treatment session will be started by the following exercises for 30 minutes as preparation for hand skill training and the second part of the session will be exercises facilitating fine motor skills a horizontal surface for one hour, Three sessions per week will last for 90 minutes, for successive Three months.
  Arms: Group (A)

SUMMARY:
The goal of this quasi-experimental study is to investigate and compare the effects of horizontal and vertical upper extremity performance on hand skills and trunk control in children with bilateral spastic cerebral palsy; could include any of the following: both gender, age ranged from 5 years to 8 years. The main question it aims to answer [is/are]:

There will be no significant difference effect between horizontal and vertical upper extremity performance on hand skills and trunk control in children with bilateral spastic cerebral palsy.

DETAILED DESCRIPTION:
This study aims to investigate the effects of to investigate and compare the effects of horizontal and vertical upper extremity performance on hand skills and trunk control in children with bilateral spastic cerebral palsy. The research will evaluate fine motor proficiency, upper extremity function and trunk stability from sitting through a controlled and structured intervention program.

Participants will undergo designed Occupational Therapy program will be applied for 90 minutes, three days per week for successive three months for the both groups by the researcher The study adopts a quasi-experimental design, with thirty participants allocated into two groups of an equal number, twenty children for each group. Two group will be identified as group (A) and group (B).

Data will be analyzed using paired t-test will be used for within group comparison before and after the intervention, for each variable and independent t-test was used to compare the demographic data and the baseline characteristics of both groups for all measured variables, pre and post treatments, with a significance level set at p < 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Children with BSCP, their chronological age will be ranged from 5 years to 8 years.
* Their level of motor function will be I or II according to Gross Motor Function Classification System - Expanded and Revised.
* The degree of spasticity for these children will ranged from grade 1 to 1⁺ according to Modified Ashworth Scale.
* Their level of fine motor function will be I or II according to The Bimanual Fine Motor Function.
* All children's level of segmental trunk control will be level 7 (full trunk control) according to Segmental Assessment of Trunk Control.
* They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

* Surgical interference in upper limbs and/or spine that may restrain the child performance during activities.
* Orthopedic problems or fixed deformities in the vertebral column and/or upper extremities.
* Uncontrolled seizures.
* Visual or hearing impairment.
* Receiving special medication affecting muscle and /or mental function.

Ages: 5 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in Fine motor proficiency | Before and after the three months of treatment
  Evaluated using the fine motor form of the Bruinink-Oseretsky test for motor proficiency 2nd edition (BOT-2)
Change in upper extremity function | Before and after the three months of treatment
  Evaluated using the Quality of Upper Extremity Skills Test (QUEST)
Change in trunk stability from sitting | Before and after the three months of treatment
  Evaluated using the Trunk Control Measurement Scale (TCMS) to assess static and anticipatory trunk control

CONTACTS AND LOCATIONS:
Overall Officials: Kamal El Sayed Shoukry, Professor Doctor, Study Chair — Department of physical therapy for growth and developmental disorder in children and its surgery, Faculty of physical therapy, Cairo University; Nanees Essam Mohamed, Professor Doctor, Study Director — Department of physical therapy for growth and developmental disorder in children and its surgery, Faculty of physical therapy, Cairo University; Gehan Mosaad Abd El-Maksoud, Professor Doctor, Study Director — Department of physical therapy for growth and developmental disorder in children and its surgery, Faculty of physical therapy, Cairo University
Locations (1):
- Faculty of physical therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No